CLINICAL TRIAL: NCT00402207
Title: The Anti-Inflammatory Effect of Extrafine HFA-Beclometasone Versus HFA-Fluticasone, by Means of Exhaled Nitric Oxide, Inflammatory Markers in Exhaled Breath Condensate and Conventional Parameters
Brief Title: The Anti-Inflammatory Effect of Extrafine HFA-Beclometasone Versus HFA-Fluticasone, by Means of Inflammometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: AstraZeneca (Industry); Teva Branded (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MEC 05-005
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2005-09

CONDITIONS: Asthma
Keywords: asthma; non-invasive inflammometry; exhaled nitric oxide; exhaled breath condensate; paediatric; extrafine HFA-beclomethasone; HFA-fluticasone
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: extrafine HFA-beclomethasone
Drug: HFA-fluticasone

SUMMARY:
Background Chronic inflammation in peripheral airways plays an important role in the pathophysiology of asthma. Extrafine hydrofluoroalkane (HFA) beclometasone is distinguished from other ICS because of its fine aerosol characteristics. As a result, there is a greater extent of deposition of extrafine HFA-beclometasone in the peripheral airways. Therefore, extrafine HFA-beclometasone may have an extra anti-inflammatory effect in children with asthma.

Aim To analyse the potential extra anti-inflammatory effect of extrafine HFA-beclometasone compared to HFA-flucticasone in children with asthma by means of alveolar nitric oxide (NO) concentration and bronchial NO flux, inflammatory markers in exhaled breath condensate (EBC), and conventional parameters.

Method In a cross-over study design of 6 months, 33 children, aged 6-12 years, with doctor diagnosed mild persistent asthma, were treated with extrafine HFA-beclometasone inhaled from an autohaler and HFA-flucticasone inhaled from a discus. Primary outcome parameters of this study were; alveolar NO concentration and bronchial NO flux. Secondary outcome parameters were inflammatory markers in EBC, lung function parameters, symptoms, presence and duration of exacerbations and adverse effects. All parameters were recorded at baseline and after each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* age 6.5 - 12 years
* children with mild-persistent asthma
* treatment with inhaled corticosteroids(≤ 500 μg HFA-Flucticasone, ≤ 800 μg Budesonide, or ≤ 800 μg HFA-Beclometasone, daily)
* allowed, but needed to be used during the entire study period;

  * short / long-acting β2-agonists
  * leukotrien receptor antagonists
  * antihistamines

Exclusion Criteria:

* Instability of asthma during the past 3 months
* Presence of a disease that may intervene with the results of this study
* Active smoking
* Mental retardation
* Inability to perform the measurements properly

Ages: 78 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33
Dates: Start 2005-08; Study Completion 2006-10

PRIMARY OUTCOMES:
status of airway inflammation after a 3 months treatment period
alveolar and bronchial exhaled nitric oxide

SECONDARY OUTCOMES:
inflammatory markers in exhaled breath condensate
lung function parameters
symptoms / symptom free days
adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte M Robroeks, MD, Principal Investigator — Maastricht University Medical Center; Rijn Jöbsis, MD, PhD, Study Director — Maastricht University Medical Center; Edward Dompeling, MD, PhD, Study Director — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands